CLINICAL TRIAL: NCT06370273
Title: Thromboprophylaxis in Lower Limb Immobilisation (TiLLI): a Multicentre Study Comprising Two Linked Open Label Phase III Randomised Controlled Trials Evaluating the Effectiveness and Cost Effectiveness of Different Methods of Pharmacological Prophylaxis for Patients With Temporary Lower Limb Immobilisation.
Brief Title: Thromboprophylaxis in Lower Limb Immobilisation
Acronym: TiLLI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1009305
Record Dates: First submitted 2024-03-21; First posted 2024-04-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Thrombosis; Injury Leg
MeSH Terms: conditions — Thrombosis; Leg Injuries | interventions — Rivaroxaban; apixaban

STUDY DESIGN:
Intervention Model Description: A pragmatic, open-label, linked pair of randomised controlled trials with common outcomes and parallel economic analysis each with internal pilot phases, conducted across 30 NHS sites
Who Masked: Outcomes Assessor
Masking Description: Open-label study. Trial Statistician and Health Economist to be blinded for analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- TiLLI-High Intervention (Active Comparator): A non-inferiority trial in people with temporary lower limb immobilisation at high risk of VTE comparing Direct Oral AntiCoagulants (DOACs) (intervention) to parenteral prophylaxis (routine care). Drug treatments will be provided for the duration of immobilisation or up to 42 days (whichever is earlier), in accordance with current NICE guidance.
  Intervention medications:
  Rivaroxaban 10mg once daily via oral ingestion. OR Apixaban 2.5mg twice daily via oral ingestion.
  Interventions: Drug: Rivaroxaban; Drug: Apixaban
- TiLLI-High Routine Care (Active Comparator): A non-inferiority trial in people with temporary lower limb immobilisation at high risk of VTE comparing Direct Oral AntiCoagulants (DOACs) (intervention) to parenteral prophylaxis (routine care). Drug treatments will be provided for the duration of immobilisation or up to 42 days (whichever is earlier), in accordance with current NICE guidance.
  Routine Care:
  Enoxaparin 40mg once daily via subcutaneous injection OR Tinzaparin 4500 IU once daily via subcutaneous injection OR Dalteparin 5000 IU once daily via subcutaneous injection OR Fondaparinux 2.5mg once daily via subcutaneous injection
  Interventions: Drug: Enoxaparin Injectable Solution; Drug: Tinzaparin Injectable Solution; Drug: Dalteparin Injectable Solution; Drug: Fondaparinux Injectable Product
- TiLLI-Low Intervention 1 (DOAC) (Active Comparator): A superiority trial in people with temporary lower limb immobilisation at low risk of VTE comparing parenteral prophylaxis (intervention) or Direct Oral AntiCoagulants (DOACs) (intervention) to no pharmacological prophylaxis (routine care). Drug treatments will be provided for the duration of immobilisation or up to 42 days (whichever is earlier), in accordance with current NICE guidance.
  Intervention medication:
  DOACs:
  Rivaroxaban 10mg once daily via oral ingestion. OR Apixaban 2.5mg twice daily via oral ingestion.
  Interventions: Drug: Rivaroxaban; Drug: Apixaban
- TiLLI-Low Intervention 2 (Parenteral prophylaxis) (Active Comparator): A superiority trial in people with temporary lower limb immobilisation at low risk of VTE comparing parenteral prophylaxis (intervention) or Direct Oral AntiCoagulants (DOACs) (intervention) to no pharmacological prophylaxis (routine care). Drug treatments will be provided for the duration of immobilisation or up to 42 days (whichever is earlier), in accordance with current NICE guidance.
  Parenteral prophylaxis:
  Enoxaparin 40mg once daily via subcutaneous injection OR Tinzaparin 4500 IU once daily via subcutaneous injection OR Dalteparin 5000 IU once daily via subcutaneous injection OR Fondaparinux 2.5mg once daily via subcutaneous injection
  Interventions: Drug: Enoxaparin Injectable Solution; Drug: Tinzaparin Injectable Solution; Drug: Dalteparin Injectable Solution; Drug: Fondaparinux Injectable Product
- TiLLI-Low Routine Care (No Intervention): A superiority trial in people with temporary lower limb immobilisation at low risk of VTE comparing parenteral prophylaxis (intervention) or Direct Oral AntiCoagulants (DOACs) (intervention) to no pharmacological prophylaxis (routine care). Drug treatments will be provided for the duration of immobilisation or up to 42 days (whichever is earlier), in accordance with current NICE guidance.
  Routine care: No pharmacological prophylaxis

INTERVENTIONS:
Drug: Rivaroxaban — 10mg once daily via oral ingestion
  Arms: TiLLI-High Intervention; TiLLI-Low Intervention 1 (DOAC)
Drug: Apixaban — 2.5mg twice daily via oral ingestion
  Arms: TiLLI-High Intervention; TiLLI-Low Intervention 1 (DOAC)
Drug: Enoxaparin Injectable Solution — 40mg once daily via subcutaneous injection
  Arms: TiLLI-High Routine Care; TiLLI-Low Intervention 2 (Parenteral prophylaxis)
Drug: Tinzaparin Injectable Solution — 4500 IU once daily via subcutaneous injection
  Arms: TiLLI-High Routine Care; TiLLI-Low Intervention 2 (Parenteral prophylaxis)
Drug: Dalteparin Injectable Solution — 5000 IU once daily via subcutaneous injection
  Arms: TiLLI-High Routine Care; TiLLI-Low Intervention 2 (Parenteral prophylaxis)
Drug: Fondaparinux Injectable Product — 2.5 mg once daily via subcutaneous injection
  Arms: TiLLI-High Routine Care; TiLLI-Low Intervention 2 (Parenteral prophylaxis)

SUMMARY:
The goal of this clinical trial is to find out the clinical and cost effectiveness of Thromboprophylaxis in participants who have been placed in a plaster cast or splint after injury.

The main questions it aims to answer are:

* whether giving tablets to people at high risks of clots after a leg injury is as good as injections (standard care)
* whether giving any medication after a leg injury is better than standard care (advice only) for people at low risk of clots.

Participants will be assessed to be high risk (TiLLI High) or low risk (TiLLI Low). People who are at high risk of clots will have either tablets or injections to reduce their risk. People at low risk will receive tablets, injections or no medication.

Drug treatments will be provided for the duration of immobilisation or up to 42 days (whichever is earlier), in accordance with current NICE guidelines. The participants will be followed up for 90 days following randomisation.

DETAILED DESCRIPTION:
People have an increased risk of blood clots when they have a leg injury treated with a plaster cast or a splint, which happens to over 70,000 people every year in the UK. Blood clots can cause long term problems in the legs and can also move to the lungs, causing serious illness and occasionally death. Medicines are available to reduce the risk of blood clots, but they can also increase the risk of bleeding. In people at high risk of clots, most hospitals use the recommended daily injections which can be uncomfortable and sometimes difficult to give. Tablets are available that reduce the risk of blood clots in other groups, but it is not known if tablets work as well as the injections for people with a leg injury. It is also not known whether people at low risk of blood clots may benefit from any medication. As such, a national research body has identified the need for further study on this topic.

The TiLLI study has two aims - to determine whether giving tablets to people at high risk of clots after a leg injury is as good as injections, and whether giving any medication is better than standard care (advice only) for people at low risk of clots.

The TiLLI study consists of two linked trials: TiLLI-High and TiLLI-Low. People who have been placed in a plaster cast or splint after a leg injury will be invited to participate. Those who agree and are at high risk of clots will enter TiLLI-High and be randomised to receive either tablets or injections to reduce their risk of blood clots; those at low risk will enter TiLLI-Low and will be randomised to receive tablets, injections, or no medication. Patients and doctors will know what medication they are taking. All patients will be provided with written guidance on the signs and symptoms of blood clots and advice on managing their medication.

Information will be collected from study participants up to 90 days after joining the study to find out whether anyone suffers blood clots or complications from the medication. This data will be collected by reviewing medical records and contacting participants as needed. To encourage people from different backgrounds to take part, the study will run from lots of different hospitals across the UK. Study materials will be translated into different languages for those who do not speak English. The investigators will collect as much information as possible from people without extra hospital visits. An independent panel will look at the data as the study progresses to decide whether it is safe to continue.

The study will cost approximately £300 per patient, which is excellent value for money. If these trials show that tablets are as effective as injections, approximately 20,000 patients will be able to avoid injections and >£1.5 million will be released back to NHS resources, every year. When the study is finished, the investigators will share the findings with staff in the NHS, patient charities and national guideline bodies. They will also publish the findings in the medical press and work with international research groups to answer further research questions on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 16 years
* Placed in temporary lower limb immobilisation (rigid cast or brace) as a result an injury that occurred within the last 7 calendar days

Exclusion Criteria:

* Hospital admission is required direct from the emergency department, minor injuries unit, or fracture clinic setting with an expected length of stay >2 calendar days.
* Absolute contraindication or known hypersensitivity to anticoagulants, including history of end stage renal failure (eGFR <20ml/min/1.73m2), hepatic failure or use of concomitant systemic treatment with azole-antimycotics (such as ketoconazole, itraconazole, voriconazole and posaconazole), HIV protease inhibitors (e.g. ritonavir) or active substances strongly inhibiting elimination pathways such as CYP3A4 or P-gp (such as clarithromycin, erythromycin or dronaderone) or a history of heparin induced thrombocytopenia.
* Pregnancy, actively seeking conception, or active breastfeeding.
* Preceding use of anticoagulant treatment for >3 calendar days at prophylactic or therapeutic dose.
* Prior enrolment in the TiLLI study.
* Non-rigid immobilisation (crepe bandage, tubigrip support, strapping).
* Time since prescription of rigid immobilisation >3 calendar days
* Co-enrolment onto a CTIMP where an anticoagulant is administered
* People lacking the capacity to consent
* Inability or refusal to use acceptable contraception up until after the last administration of IMP. Only applicable for women of childbearing potential who have been randomised to receive apixaban or rivaroxaban

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10044 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite of net clinical benefit comprising clinical VTE event, major bleeding, and cause-specific mortality | Within 90 days of randomisation
  To estimate and draw inferences on the difference in a composite outcome of net clinical benefit between treatment groups. A composite primary outcome of net clinical benefit, comprising symptomatic VTE events (any deep vein thrombosis or pulmonary embolism), major bleeding or cause-specific mortality (death from either pulmonary embolus or major bleeding) used as a binary variable ('1' is any event occurred, '0' if none of the events occurred).

SECONDARY OUTCOMES:
Symptomatic VTE event occurrence | Within 90 days from randomisation
  To compare symptomatic VTE events (any deep vein thrombosis or pulmonary embolism) (an individual component of primary composite outcome) between treatment groups as a binary variable ('1' if any event occurred, '0' if no event occurred). Symptomatic VTE events objectively defined by ISTH criteria.
Major bleeding occurrence | Within 42 days from randomisation
  To compare major bleeding events (an individual component of primary composite outcome) between treatment groups as a binary variable ('1' if any event occurred, '0' if no event occurred). Major bleeding events objectively defined by ISTH criteria.
Cause-specific mortality occurrence | Within 90 days from randomisation
  To compare cause-specific mortality events (an individual component of primary composite outcome) between treatment groups as a binary variable ('1' if any event occurred, '0' if no event occurred).
Adverse and Serious adverse events | Within 90 days from randomisation.
  To estimate and draw inferences on the difference in complications (including clinically relevant non-major bleeding and surgical site bleeding) objectively defined by ISTH criteria, between treatment groups.
Medication adherence | Up to 42 days from randomisation
  To report participant adherence to allocated anticoagulant verified through digital response system.
Health utility (EQ-5D-5L) | Up to 90 days post randomisation.
  To estimate and draw inferences on differences in quality-of-life measures between treatment groups. Using the EuroQol 5 Dimensions 5 Level (EQ-5D-5L), a validated instrument comprising a self-rated health VAS and a five-domain health status questionnaire related to daily activities. Will collect for 4 timepoints: pre injury (completed retrospectively within 7 days following randomisation), 7 days following randomisation, 42 days following randomisation, and 90 days following randomisation
Patient satisfaction regarding the burdens and benefits of anticoagulation | Collected within 42 days following randomisation when the participants stops study treatment.
  To estimate and draw inferences on the acceptability of different prophylactic anticoagulants using the validated Anti Clot Treatment Scale (ACTS) for patients allocated to drug treatments. The scale is a 15-item patient-reported instrument of satisfaction with anticoagulation treatment, with separate internal measures of burden and benefits.
Hospital readmission/reattendance | Within the first 90 days.
  To estimate and draw inferences on the difference in resource use (including hospital readmission/reattendance), cost, quality of life-adjusted survival and relative cost effectiveness between treatment groups. Using bespoke Case Report Forms and review of EHR, research staff to collect information on resources required to deliver subsequent care reviews (including scheduled clinic and unscheduled hospital attendance), and investigations.
Health and social care resource use | Within the first 90 days
  To estimate the health and social care resource use and costs and the relative cost effectiveness between treatment groups. Using bespoke Case Report Forms and review of EHR, research staff to collect information on health and social care resource use.
Patient longer term outcome VTE and bleeding data | Informed by directly measured events up to 90 days.
  To estimate longer term outcomes, such as post thrombotic syndrome, chronic thromboembolic pulmonary hypertension and bleeding complications and draw inferences on cost effectiveness, by using an existing VTE model with risk-adjusted, population specific effect estimates from this study. This will allow efficient, value for money inferences to made about long-term sequelae of VTE events and determine whether detailed long-term follow-up of participants would be worthwhile. Clinically relevant non-major bleeding events, major bleeding events and symptomatic bleeding events objectively defined by ISTH criteria.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton, Surrey
  - Barts Health NHS Trust, London
  - Northern Care Alliance NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No